CLINICAL TRIAL: NCT05332119
Title: Effectiveness of Virtual Reality on Pain and Anxiety During the Removal of Chest Drains in Critically-ill Patients
Brief Title: Virtual Reality During the Removal of Chest Drains in Critically-ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gemma Via Clavero (Other)
Responsible Party: Sponsor-Investigator, Gemma Via Clavero, PhD. Advanced Practice Critical Care Nurse, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICPS001/22
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Pain; Anxiety
Keywords: Virtual reality glasses
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Each patient will be randomized in a 1:1 ratio between the two arms of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): The intervention will consist of the use of VR glasses during the removal of chest drains. The VR content has been developed by VR Pharma Immersive Technologies (LtD). Its main objective is to improve patient experience and have better management of pain and anxiety. Chest drains are removed following the usual protocol.
  Interventions: Device: VR glasses
- Control group (Sham Comparator): Patients in the control group will be cared for with the usual care protocol.
  Interventions: Other: Control group

INTERVENTIONS:
Device: VR glasses — Patients will watch a virtual world in VR glasses during the painful procedure. They will be able to choose between 3 VR content based on their preferences.
  Arms: Virtual reality
Other: Control group — Patients will not receive distraction during chest drain removal
  Arms: Control group

SUMMARY:
Appropriate pain and anxiety management of critically-ill patients during bedside procedures remains a big challenge. Clinical Practice Guidelines recommend preemptive analgesia or non-pharmacological interventions, such as relaxation techniques or distraction, to prevent and treat pain during nursing procedures. One of the most painful procedures in the Intensive Care Unit (ICU) is the removal of chest drains in post-cardiac surgical patients.

Virtual reality (VR) is a computer-generated simulation of a 360º immersive world in which the patient can receive visual and auditory stimuli that distract them from the real environment. Current research has demonstrated that VR reduced pain and anxiety in intravenous catheter insertions or wound care.

The primary objective of the study is to evaluate the effectiveness of VR on pain and anxiety during the removal of chest drains, in post-cardiac surgical patients. The hypothesis is that VR reduces both pain and anxiety, in critically-ill patients, during the removal of chest drains in post-cardiac surgical patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, prospective study of two parallel groups of patients during the removal of chest drains:

Group 1: removal of chest drains according to the usual management protocol.

Group 2: removal of chest drains according to the usual management protocol supplemented by the use of virtual reality glasses (VR glasses)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients with Richmond Agitation-Sedation Scale (RASS) between -1 to RASS +1
* Patients undergoing cardiac surgery
* Patients with chest drains
* Patients who voluntarily agree to participate (informed consent form)

Exclusion Criteria:

* Patients with a language barrier
* Patients with cognitive impairments
* Patients with neuromuscular blockers
* Patients with a previous history of documented anxiety
* Patients with epilepsy
* Hemodynamically unstable patients
* Face or ocular infections, with could contaminate VR glasses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Procedural pain score | Baseline
  Numerical rating scale (NRS). The pain can be scored from 0 to 10 (0=no pain, 10= worst possible pain)
Procedural pain score | 1 minute after the removal of chest drains
  Numerical rating scale (NRS). The pain can be scored from 0 to 10 (0=no pain, 10= worst possible pain)
Procedural pain score | 30 minutes after the removal of chest drains
  Numerical rating scale (NRS). The pain can be scored from 0 to 10 (0=no pain, 10= worst possible pain)
Procedural anxiety score | Baseline
  State-Trait Anxiety Inventory (STAI scale)- trait state. The anxiety can be scored from 0 to 60 (0=no anxiety, 60=worst possible anxiety)
Procedural anxiety score | 1 minute after the removal of chest drains
  State-Trait Anxiety Inventory (STAI scale)- trait state. The anxisety can be scored from 0 to 60 (0=no anxiety, 60=worst possible anxiety)
Procedural anxiety score | 30 minutes after the removal of chest drains
  State-Trait Anxiety Inventory (STAI scale)- trait state. The anxisety can be scored from 0 to 60 (0=no anxiety, 60=worst possible anxiety)

SECONDARY OUTCOMES:
Sociodemographic and clinical factors | Baseline
  Age, gender, past medical history
Blood pressure | Baseline
  Systolic, Diastolic and mean blood pressure measure in mmHg
Blood pressure | 1 minute after the removal of chest drains
  Systolic, Diastolic and mean blood pressure measure in mmHg
Blood pressure | 30 minutes after the removal of chest drains
  Number of systolic, diastolic and mean blood pressure measure in mmHg
Heart rate | Baseline
  Number in beats per minute
Heart rate | 1minute after the removal of chest drains
  Number in beats per minute
Heart rate | 30 minutes after the removal of chest drains
  Number in beats per minute
Respiratory rate | Baseline
  Number in breaths per minute
Respiratory rate | 1 minute after the removal of chest drains
  Number in breaths per minute
Respiratory rate | 30 minutes after the removal of chest drains
  Number in breaths per minute
Type of cardiac surgery | Baseline
  Type
Type of chest drains | At baseline
  Mediastinal or pleural drains
Number of chest drains | At baseline
  Number
Dose of analgesic drugs | 1 hour before the procedure
  Cumulated dose of analgesia drugs
Patient satisfaction | 30 minutes
  Numerical Rating Scale (NRS). Patient's satisfaction will be scored from 0 to 4 (0= unsatisfied, 4=very satisfied).
Adverse events | 30 minutes
  Type of adverse events experienced by patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Nordness MF, Hayhurst CJ, Pandharipande P. Current Perspectives on the Assessment and Management of Pain in the Intensive Care Unit. J Pain Res. 2021 Jun 14;14:1733-1744. doi: 10.2147/JPR.S256406. eCollection 2021. PMID 34163231
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Sadeghi AH, Mathari SE, Abjigitova D, Maat APWM, Taverne YJHJ, Bogers AJJC, Mahtab EAF. Current and Future Applications of Virtual, Augmented, and Mixed Reality in Cardiothoracic Surgery. Ann Thorac Surg. 2022 Feb;113(2):681-691. doi: 10.1016/j.athoracsur.2020.11.030. Epub 2020 Dec 19. PMID 33347848
- [Background] Ioannou A, Papastavrou E, Avraamides MN, Charalambous A. Virtual Reality and Symptoms Management of Anxiety, Depression, Fatigue, and Pain: A Systematic Review. SAGE Open Nurs. 2020 Aug 27;6:2377960820936163. doi: 10.1177/2377960820936163. eCollection 2020 Jan-Dec. PMID 33415290